CLINICAL TRIAL: NCT03725267
Title: Melatonin for Renal Protection in Patients Receiving Polymyxin B:a Randomized Clinical Trial
Brief Title: Melatonin for Renal Protection in Patients Receiving Polymyxin B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to COVID 19 pandemic social isolation measures, we had to stop recruting hospitalized patients.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 77374017.1.0000.5327
Record Dates: First submitted 2018-10-11; First posted 2018-10-31 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Acute Kidney Injury; Melatonin; Polymyxin B Adverse Reaction
Keywords: Melatonin; Polymixin B; RIFLE; Nephrotoxicity
MeSH Terms: conditions — Acute Kidney Injury | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo-controlled, 2-arm parallel trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Melatonin and placebo pills will be manipulated in identical format. The pharmacist will provide similar packets of 7 pills each numbered from 1 to 100. Each packet will have placebo or melatonin according to a randomization list previously sent from a researcher responsible (not involved with intervention). Patients will be consecutively enrolled and receive the packet following the order of one to 100.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Patients will receive 1 pill each day with 30 mg of Melatonin during polymyxin B treatment for a maximum of 14 days.
  Interventions: Drug: Melatonin Pill
- Placebo (Placebo Comparator): Patients will receive 1 pill each day with Placebo during polymyxin B treatment for a maximum of 14 days.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Melatonin Pill — Patients will receive 1 pill of melatonin each day during polymyxin B therapy for a maximum of 14 days.
  Arms: Melatonin
Drug: Placebo oral capsule — Patients will receive 1 pill of placebo each day during polymyxin B therapy for a maximum of 14 days.
  Arms: Placebo

SUMMARY:
This study has the objective to evaluate the effect in renal function of 30mg of Melatonin versus placebo in patients ≥18 years old treated with polymyxin B. The development of nephrotoxicity will be evaluated by RIFLE(Risk, Injury, Failure, Loss, End stage renal disease) score and KIM-1 urinary biomarker for the first 14 days of polymyxin B therapy.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo controlled, phase 2 superiority trial.

Patients ≥18 years old admitted in two tertiary care hospitals from Porto Alegre-Brazil receiving intravenous polymyxin B (PMB) will be included after agreeing with the informed consent. Exclusion criteria will be use of PMB for less than 48 hours, chronic dialysis or glomerular filtration rate <10ml/min or Intensive Care Unit (ICU) admission at baseline, previous regular use of melatonin, pregnancy, unability to receive oral medications or deprived from liberty individuals. All eligible patients will be consecutively recruited.

Primary outcome will be nephrotoxicity evaluated by RIFLE criteria. Secondary outcomes will be development of Renal Failure (by RIFLE criteria), Kidney Injury Molecule-1 (KIM-1) urinary biomarker evaluated at days 2,4 and 7 after the start of PMB and 30 day mortality. Potential confounding factors will be evaluated, such as: demographic variables, comorbidities, PMB dose, concomitant use of other antimicrobials, though concentration of PMB after the 4th dose of the antibiotic.

Patients will be randomized in a 1:1 ratio by a computer system in blocks of 4 for melatonin 30mg or placebo. Analysis will be stratified by center. Patients, attending physicians and researchers responsible for the intervention and data collection will be blinded.

Univariate analysis of variables that could potentially impact on nephrotoxicity will be done by T-test or Wilcoxon rank-sum and Fisher test according to the variables characteristics. A Cox regression model for time to nephrotoxicity during PMB therapy will be done, censoring patients if death, end of therapy or completion of 14 days of PMB therapy. The main analysis will be for intention- to-treat and a secondary per-protocol analysis will be done for patients that received at least 80% of the planned doses. All tests will be two-sided and P≤0.05 will be considered statistically significant.

A subgroup analysis is planned for patients with baseline glomerular filtration rate ≥60ml/min and ≥60years old.

The calculated sample size for this study is of 100 patients, 50 in each arm. An interim analysis is planned when half of the sample is recruited (25 in each arm). If the number of patients that achieve nephrotoxicity criteria is at least 30% less in one of the arms compared to the other, with a P≤0,01, the study will be interrupted.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment with polymyxin B ( a second inclusion will be accepted if the end of the previous treatment was more than 30-days before enrollment)
2. Agreement with the consent form

Exclusion Criteria:

1. Suspension of polymyxin B therapy with <48hs
2. Death in <48hs
3. Dialysis or Glomerular Filtration Rate (GFR) <10 ml/min at the beginning of treatment by the Modification in Diet in Renal Disease (MDRD) formula
4. Lactose intolerance
5. ICU admission at the beginning of therapy
6. Previous regular use of Melatonin
7. Pregnancy
8. Patients deprived from liberty
9. Unability to receive oral medication (i.e total parenteral nutrition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury according to RIFLE criteria | 14 days Renal Failure.
  Acute Kidney Injury measured by Risk, Injury, Failure, Loss and End Stage Renal Disease (RIFLE) score, which takes in account variations of creatinin levels and glomerular filtration rate compared to baseline values: Risk (R) increase in 1.5 times the creatinine value or decrease >25% glomerular filtration rate; Injury (I) increase in 2.0 times the creatinine value or decrease >50% glomerular filtration rate, Failure (F) increase in 3.0 times the creatinine value or decrease >75% glomerular filtration rate. Due to the study follow-up time we won´t be able to evaluate Loss (L) nor End Stage Renal Disease (E)- which would require at least 4 weeks of renal function monitoring ( we will follow patients only during polymyxin B treatment, up to 14 days).The better outcome would be not fulfilling any RIFLE criteria and the worse outcome would be Failure (F).

SECONDARY OUTCOMES:
Renal Failure according to RIFLE criteria | 14 days
  Renal failure by RIFLE criteria is considered and increase of 3 times the creatinin values compared to baseline or a decrease of 75% of the glomerular filtration rate.
Kidney Injury Molecule-1 (KIM_1) | 7 days
  Urinary biomarker measured on days 2, 4 and 7 after the beginning of PMB therapy. The rise in the biomarker values (days 4 and 7) compared to baseline (day 2)will be an early measure of kidney injury.
30-day mortality | 30 days
  All cause mortality after 30-days of the beginning of PMB therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena P Rigatto, Professor, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Pontificia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided
We will provide individual participant data if required by direct contact with our PI.